CLINICAL TRIAL: NCT04885322
Title: Effects of PFC tDCS on Cognitive Control, Attention Lapses and Coordinated Neural Activity in the Theta and Alpha Bands
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1344169-8
Record Dates: First submitted 2021-05-04; First posted 2021-05-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- DLPFC Stimulation (Experimental): Intervention. 20 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Occipital Stimulation (Experimental): Intervention. 20 minutes of 2 mA direct current stimulation over the occipital cortex.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham Stimulation (Sham Comparator): Placebo Comparator. 0.5-1 minutes of 2 mA direct current stimulation over the dorsolateral prefrontal cortex followed by 19-19.5 minutes of sham stimulation
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — In tDCS, saline-soaked electrodes are temporary affixed to the scalp and connected to a battery-powered current generator. A weak (2 mA) constant current is then briefly applied (~20 minutes) to stimulate the targeted brain area. The targeted brain area is determined by the Study Arm.

SUMMARY:
The purpose of this study is to better understand the neural correlates of higher-order cognition, both in the healthy brain and in schizophrenia, and to determine how these mechanisms are modulated by transcranial direct current stimulation (tDCS) at frontal and occipital scalp sites. Testing the effects of tDCS at these scalp sites on cognitive task performance will help us understand the roles of the brain regions corresponding to these sites during higher-order cognitive processing (language comprehension, cognitive control, and related attention and memory processes). Behavioral and electrophysiological (EEG) measures will be used to assess cognitive performance. Our overarching hypothesis is that stimulating prefrontal circuits with tDCS can improve cognitive control performance, and ultimately performance on a range of cognitive tasks, as compared to stimulating a different cortical region (occipital cortex) or using sham stimulation.

This study is solely intended as basic research in order to understand brain function in healthy individuals and individuals with schizophrenia. This study is not intended to diagnose, cure or treat schizophrenia or any other disease.

ELIGIBILITY:
Inclusion Criteria:

* between ages of 18 and 50
* ability to sufficiently speak and understand English so as to be able to understand and complete cognitive tasks
* ability to give valid informed consent

Exclusion Criteria:

* no history of head trauma
* no current or previous history of treatment with psychotropic medication
* corrected vision 20/30 or better
* tDCS/MRI contraindications, including: pregnancy, ferrous metal in any part of the body, serious medical conditions, claustrophobia, metallic implants, skin damage, conditions such as eczema at electrode sites, cranial pathologies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Behavioral Cognitive Control Measures on the Stroop Task | Through study completion, an average of 1 month
  Incongruent versus Congruent difference in error rate and reaction time
EEG Cognitive Control Measures on the Stroop Task | Through study completion, an average of 1 month
  response-locked power in the theta frequency band (4-7 Hz)
Behavioral Attention Lapse Measures on the Stroop Task | Through study completion, an average of 1 month
  Error Rate on Incorrect Congruent trials (Full Lapses) and Slow-but-Correct Congruent trials (Partial Lapses)
EEG Attention Lapse Measures on the Stroop Task EEG Attention Lapse Measures on the Stroop Task | Through study completion, an average of 1 month
  Pre-trial power in the alpha frequency band (8-12 Hz)
Behavioral Cognitive Control Measures on the Change Detection Task Behavioral Cognitive Control Measures on the Change Detection Task | Through study completion, an average of 1 month
  WM storage capacity (k-max)
EEG Cognitive Control Measures on the Change Detection Task | Through study completion, an average of 1 month
  delay period power in the theta frequency band (4-7 Hz)
Behavioral Attention Lapse Measures on the Change Detection Task | Through study completion, an average of 1 month
  Attention factor (a); Guess factor (g)
EEG Attention Lapse Measures on the Change Detection Task | Through study completion, an average of 1 month
  Pre-trial power in the alpha frequency band (8-12 Hz)
Delivered tDCS Dose to PFC | Through study completion, an average of 1 month
  Estimated electric field in PFC region of interest

CONTACTS AND LOCATIONS:
Locations (1):
- Imaging Research Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No